CLINICAL TRIAL: NCT05433480
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Compare Fulvestrant Plus BPI-16350 or Plus Placebo in Patients With HR+, HER2- Locally Advanced, Recurrent or Metastatic Breast Cancer With Disease Progression Following Endocrine Therapy
Brief Title: A Study of BPI-16350 in Combination With Fulvestrant in Patients With HR+ and HER2- Locally Advanced, Recurrent or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTP-66732
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Intervention Drug: BPI-16350, Fulvestrant
  Interventions: Drug: BPI-16350; Drug: Fulvestrant
- control group (Placebo Comparator): Intervention Drug: Placebo, Fulvestrant
  Interventions: Drug: placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: BPI-16350 — BPI-16350 400 mg, orally once daily
  Arms: experimental group
Drug: placebo — Placebo 400 mg, orally once daily
  Arms: control group
Drug: Fulvestrant — Fulvestrant 500 mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 for every cycle until progressive disease

SUMMARY:
This is a phase III clinical trial to evaluate the efficacy and safety of BPI-16350 in combination with Fulvestrant versus placebo combined with Fulvesrant in Patients who have HR positive and HER2 negative locally advanced，recurrent or metastatic breast cancer with disease progression following endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has the pathologically-confirmed diagnosis of locally advanced, recurrent or metastatic, HR positive, HER2 negative Breast Cancer
* One previous line of chemotherapy for advanced/metastatic disease is allowed
* Disease Progression following endocrine therapy
* Have postmenopausal status
* Have 1 of the following, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1: measurable disease or nonmeasurable bone-only disease
* ECOG: 0~1
* Adequate organ function

Exclusion Criteria:

* Previous treatment with cytotoxic drugs within 4 weeks before enrollment
* Previous treatment with endocrine or small molecule drug tyrosine kinase inhibitor TKI within 2 weeks before enrollment
* Patients who received prior treatment with any CDK4/6 inhibitor, everolimus or fulvestant
* HER2 positive
* Patients with major surgery within 4 weeks, severe or unstable systemic disease, unstable/symptomatic CNS metastasis, other malignant tumors, ILD, clinical significant cardiac disease, bleeding or embolic disease, active infectious disease, conditions affecting drug swallow and absorption, etc
* Pregnancy or lactation
* Other conditions considered not appropriate to participate in this trial by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed PFS | up to 3 years
  The PFS time is measured from the date of randomization to the date of objective progression or the date of death due to any cause, whichever is earlier.

SECONDARY OUTCOMES:
IREC-assessed PFS | up to 3 years
  The PFS time is measured from the date of randomization to the date of objective progression or the date of death due to any cause, whichever is earlier.
ORR | up to 3 years
  The proportion of patients with CR or PR according to RECIST v1.1
DCR | up to 3 years
  The proportion of patients with CR, PR, or SD according to RECIST v1.1
DOR | up to 3 years
  The time from the date of first evidence of a CR or PR to the date of objective progression or death from any cause, whichever is earlier
CBR | up to 3 years
  The proportion of patients with CR, PR, or SD ≥6 months according to RECIST v1.1
OS | up to 5 years
  The time from the date of randomization to the date of death from any cause
AEs and SAEs | up to 3 years
  Number of Participants With adverse events (AEs) and serious adverse events (SAEs) Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0
EORTC QLQ-C30 | up to 5 years
  Changes in scores from baseline using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)
Evaluate the pharmacokinetics of BPI-16350 | Up to 3 cycles(each cycle is 28 days)
  Based on blood plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Ph.D, Principal Investigator — Fudan University; Shuseng Wang, Principal Investigator — Sun Yat-Sen University Cancer Hospital
Locations (64):
- China (64):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Medical Center of the PLA General Hospital, Beijing, Beijing Municipality
  - The Seventh Medical Center of the PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Ximen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Hospital, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cangzhou Hospital of Integrated TCM-WM·Hebei, Cangzhou, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The first Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Fifth Hospital in WuHan, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The First People's Hospital Of Changde City, Changde, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Loudi Central Hospital, Loudi, Hunan
  - Shaoyang Central Hospital, Shaoyang, Hunan
  - Yongzhou Central Hospital, Yongzhou, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Jilin Hospital of Chinese Literature, Siping, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital ＆ Institute, Shenyang, Liaoning
  - Inner Mongolia People's Hospital, Hohhot, Neimenggu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Weifang People's Hospital, Weifang, Shangdong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital&Institute, Chengdu, Sichuan
  - The Sixth People's Hospital of Chengdu, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tao Z, Zhang J, Zheng Q, Wang Y, Cai L, Xu H, Xu X, Kong X, Ding S, Hao C, Wang H, Zong H, Jin X, Wang X, Li Y, Yang X, Li W, Du X, Chen H, Wu P, Li P, Mao L, Ding L, Hu X, Wang S. Tibremciclib or Placebo Plus Fulvestrant in Hormone Receptor-Positive and ERBB2-Negative Advanced Breast Cancer After Endocrine Therapy: A Randomized Clinical Trial. JAMA Oncol. 2025 Sep 1;11(9):1055-1063. doi: 10.1001/jamaoncol.2025.2092. PMID 40742733
- [Derived] Zhang J, Liu R, Gao S, Chen W, Han X, Wang Z, Zhou H, Wang Y, Chen J, Ma Y, Liu K, Shen Z, Ding L, Li P, Hu X. A phase I dose-escalation and dose-expansion study of tibremciclib, a novel CDK4/6 inhibitor, monotherapy and in combination with fulvestrant in HR-positive/HER2-negative advanced breast cancer. ESMO Open. 2025 Jun;10(6):105121. doi: 10.1016/j.esmoop.2025.105121. Epub 2025 May 21. PMID 40403388